CLINICAL TRIAL: NCT06365580
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Single and Multiple Ascending Doses of Kylo-0603 Capsules in Healthy Subjects
Brief Title: Dose Escalation Study of Kylo-0603 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kylonova (Xiamen) Biopharma co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kylo-0603-I-C01
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-04

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kylo-0603 (Experimental): In part 1, subjects will receive single dose Kylo-0603 orally at dose levels of 0.3 mg, 0.6 mg, 1.2 mg, 2.4 mg, 4.6 mg, 8.6 mg, 12 mg, 16 mg and 20 mg on Day 1. In part 2, subjects will receive Kylo-0603 4.6 mg on Day 1 in fasted state and on Day 4 after a standard high-fat meal. In part 3, subject will receive Kylo-0603 orally once daily for 14 days at dose levels of 1.2 mg, 2 mg, 4 mg, 8 mg, 12 mg, and 16 mg.
  Interventions: Drug: Kylo-0603 capsule
- Placebo (Placebo Comparator): Subjects will receive matching placebo in part 1, part 2 and part 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kylo-0603 capsule — Administrated orally.
  Arms: Kylo-0603
Drug: Placebo — Administrated orally.
  Arms: Placebo

SUMMARY:
This clinical trial is the first-in-human study of Kylo-0603. The purpose of this randomized, double-blind, placebo-controlled phase 1 study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and effect of food of Kylo-0603 in healthy Chinese adult subjects.

DETAILED DESCRIPTION:
The study consists of three parts: single ascending doses (Part 1), food effect (Part 2) and multiple ascending doses (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 55 years old, inclusive;
* Body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive；
* Having no clinically significant disorder, condition or disease at screening and before first dosing;
* Female subjects must not be able to get pregnant and male subjects must agree to adhere to contraception restrictions;
* Willing to comply with protocol required visits and assessments, and provide written informed consent.

Exclusion Criteria:

* History of cardiovascular, respiratory, digestive, liver, urinary, hematological, endocrine, metabolic, immune, cutaneous, or psychoneurotic diseases；
* History of evidence of malignant tumor or Gilbert syndrome;
* Positive screen of Hepatitis B surface antigen, hepatitis C virus, human immunodeficiency virus or syphilis infection;
* History of tuberculosis infection;
* History of alcohol abuse within 12 months before dosing;
* History of drug abuse within 3 months before screening;
* History of blood donations or blood loss of 400 ml and more within 3 months before dosing;
* Pregnant or breast-feeding women;
* Other exclusion criteria applied per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events | up to 3 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter of maximum observed concentration (Cmax) | up to 3 weeks
PK parameter of time of maximum observed concentration (Tmax) | up to 3 weeks
PK parameter of area under the concentration time curve (AUC) | up to 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China